CLINICAL TRIAL: NCT00650156
Title: A Randomized, Parallel-group, Open-Label, Pharmacokinetic and Safety Study With Adalimumab in Chinese Subjects With Mild Rheumatoid Arthritis.
Brief Title: Pharmacokinetic and Safety Study With Adalimumab in Chinese Subjects With Mild Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Beverly Paperiello, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-017
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2010-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 mg adalimumab (Experimental)
  Interventions: Biological: adalimumab
- 80 mg Adalimumab (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg single sc dose
  Other Names: ABT-D2E7; Humira
  Arms: 40 mg adalimumab
Biological: adalimumab — 80 mg single sc dose
  Other Names: ABT-D2E7; Humira
  Arms: 80 mg Adalimumab

SUMMARY:
Pharmacokinetic and Safety Study with Adalimumab in Chinese Subjects with Mild Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ages 18 years and older.
* Mild RA.
* Body weight less than 100 kg.

Exclusion Criteria:

* Wheelchair-bound or bedridden.
* Joint surgery involving joints to be assessed within this study, within two months prior to the Screening visit.
* Intra-articular, intramuscular or intravenous (IV) administration of corticosteroids within 28 days prior to the Screening visit.
* Prior treatment with any TNF antagonist, including adalimumab.
* Positive tuberculin PPD 5.
* Female subjects who are pregnant or breast-feeding.
* History of HIV or of being immuno-compromised.
* History of malignancy.
* Poorly controlled medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of a single subcutaneous dose of 40 and 80 mg adalimumab | Days 1, 2, 4, 6, 8, 11, 15, 22, & 29

SECONDARY OUTCOMES:
Adverse event profile | follow up to day 70 after dose
VAS assessments | Days 1, 15 and 29
Swollen and Tender Joint counts | Days 1, 15 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 7181, Shanghai, China

REFERENCES:
- [Background] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778